CLINICAL TRIAL: NCT03517969
Title: A Phase 2 Study of M6620 (VX-970, Berzosertib) in Combination With Carboplatin Compared With Docetaxel in Combination With Carboplatin in Metastatic Castration-Resistant Prostate Cancer
Brief Title: M6620 and Carboplatin With or Without Docetaxel in Treating Patients With Metastatic Castration-Resistant Prostate Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2018-00790; NCI-2018-00790 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 10191 (Other: Dana-Farber - Harvard Cancer Center LAO); 10191 (Other: CTEP); UM1CA186709 (NIH)
Record Dates: First submitted 2018-05-07; First posted 2018-05-08 (Actual); Results first posted 2025-05-08 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-10

CONDITIONS: Castration-Resistant Prostate Carcinoma; Metastatic Prostate Carcinoma; Stage IV Prostate Cancer AJCC v8
MeSH Terms: conditions — Prostatic Neoplasms | interventions — berzosertib; Carboplatin; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A (docetaxel, carboplatin) (Active Comparator): Patients receive docetaxel IV over 60 minutes and carboplatin IV over 30 minutes, or carboplatin alone on day 1. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity. Patients who have PSA progression or radiographic progression may crossover to Arm B.
  Interventions: Drug: Carboplatin; Drug: Docetaxel; Other: Laboratory Biomarker Analysis
- Arm B (carboplatin, berzosertib) (Experimental): Patients receive carboplatin IV over 30 minutes on day 1 and berzosertib IV over 60-90 minutes on days 2 and 9. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Berzosertib; Drug: Carboplatin; Other: Laboratory Biomarker Analysis

INTERVENTIONS:
Drug: Berzosertib — Given IV
  Other Names: 2-Pyrazinamine, 3-(3-(4-((Methylamino)methyl)phenyl)-5-isoxazolyl)-5-(4-((1-methylethyl)sulfonyl)phenyl)-; M 6620; M6620; VX 970; VX-970; VX970
  Arms: Arm B (carboplatin, berzosertib)
Drug: Carboplatin — Given IV
  Other Names: Blastocarb; Carboplat; Carboplatin Hexal; Carboplatino; Carboplatinum; Carbosin; Carbosol; Carbotec; CBDCA; Displata; Ercar; JM-8; JM8; Nealorin; Novoplatinum; Paraplatin; Paraplatin AQ; Paraplatine; Platinwas; Ribocarbo
Drug: Docetaxel — Given IV
  Other Names: Docecad; RP 56976; RP-56976; RP56976; Taxotere; Taxotere Injection Concentrate
  Arms: Arm A (docetaxel, carboplatin)
Other: Laboratory Biomarker Analysis — Correlative studies

SUMMARY:
This phase II trial studies how well berzosertib (M6620) and carboplatin with or without docetaxel works in treating patients with castration-resistant prostate cancer that has spread to other places in the body (metastatic). M6620 may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Drugs used in chemotherapy, such as carboplatin and docetaxel, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Giving M6620, carboplatin and docetaxel may work better in treating patients with metastatic castration-resistant prostate cancer compared to carboplatin and docetaxel alone.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To assess the difference in response rate (either achievement of prostate specific antigen [PSA] reduction of greater than 50% or radiographic response by Response Evaluation Criteria in Solid Tumors [RECIST] 1.1) of the combination of berzosertib (M6620) (VX-970, berzosertib) and carboplatin as compared to the combination of docetaxel and carboplatin.

SECONDARY OBJECTIVES:

I. To assess the difference in time to PSA progression by Prostate Cancer Working Group (PCWG)2 criteria of the combination of M6620 (VX-970, berzosertib) and carboplatin as compared to the combination of docetaxel and carboplatin.

II. To describe radiographic progression-free survival and progression-free survival by PCWG3 criteria in both arms of the study.

III. Assess the relationship with homologous recombination deficiency (HRD) detected from baseline tumor biopsy with response to the combination of M6620 (VX-970, berzosertib) and carboplatin and the combination of docetaxel and carboplatin.

IV. To describe the safety and adverse events from the combination of M6620 (VX-970, berzosertib) + carboplatin as well the combination of docetaxel + carboplatin.

EXPLORATORY OBJECTIVES:

I. Comparison of overall survival in the two arms of the study. II. Explore response rate, time to PSA progression, radiographic progression-free survival, and progression-free survival by PCWG3 criteria in patients who initially receive docetaxel + carboplatin after crossover to M6620 + carboplatin.

III. To assess the relationship with homologous recombination deficiency (HRD) detected from baseline circulating free deoxyribonucleic acid (DNA) (cfDNA) with response to the combination of M6620 and carboplatin and the combination of docetaxel and carboplatin, and describe alterations seen in cfDNA (and optional tumor biopsy) at end of study.

OUTLINE: Patients are randomized to 1 of 2 groups.

ARM A (docetaxel, carboplatin): Patients receive docetaxel intravenously (IV) over 60 minutes and carboplatin IV over 30 minutes on day 1 or carboplatin alone on day 1. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity. Patients have PSA progression or radiographic progression may crossover to Arm B.

ARM B (carboplatin, berzosertib): Patients receive carboplatin IV over 30 minutes on day 1 and berzosertib IV over 60-90 minutes on days 2 and 9. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up between 30-42 days.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have histologically or cytologically confirmed prostate cancer (code 10036910) with progressive disease at the time of study entry by either

  * Sequence of at least 2 rising PSA values at a minimum of 1-week intervals
  * Radiographic progression per RECIST1.1 for soft tissue and/or per PCWG3^2 for bone, with or without PSA progression
* Patients must have metastatic disease by bone scan or other nodal or visceral lesions on computed tomography (CT) or magnetic resonance imaging (MRI) and a castrate level of testosterone (< 50 ng/dL) and evaluable for disease response by either

  * Baseline PSA >= 2.0 ng/mL OR
  * Measurable disease per RECIST 1.1
  * NOTE: Subjects must maintain a castrate state; if they have not had an orchiectomy, they must continue to receive luteinizing hormone-releasing hormone (LHRH) or gonadotropin-releasing hormone (GnRH) agonists or antagonists unless intolerant
* At least 2 prior treatments for castration resistant prostate cancer as follows:

  * Past progression or intolerance to at least one secondary hormonal therapy (abiraterone, enzalutamide, galeterone, apalutamide, darolutamide, orteronel, seviteronel or equivalent)
  * Past progression or intolerance to taxane-based chemotherapy
* Eastern Cooperative Oncology Group (ECOG) performance status =< 1 (Karnofsky >= 70%)
* Leukocytes >= 3,000/mcL
* Absolute neutrophil count >= 1,500/mcL
* Hemoglobin >= 9 g/dL (transfusion permitted)
* Platelets >= 150,000/mcL (without transfusion or growth factor in prior 28 days)
* Total bilirubin =< 1.5 x institutional upper limit of normal, unless the subject has known or suspected Gilbert's syndrome
* Aspartate aminotransferase (AST) (serum glutamic-oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 2.5 x institutional upper limit of normal or =< 5 x if presence of liver metastases
* Creatinine clearance >= 40 mL/min/1.73 m^2
* Prior treatment with mTOR inhibitors, cytostatic tyrosine kinase inhibitor (TKI), or biologic therapies allowed
* Prior treatment with PARP inhibitors permitted
* Patients with allergy or intolerance to docetaxel, grade 2 neuropathy are allowed on study, but if randomized to Arm A will receive carboplatin as a single agent (area under curve [AUC] 5) rather than docetaxel+carboplatin; they must be fit for carboplatin chemotherapy as determined by the treating investigator
* Presence of a lesion (bone or soft tissue) amenable to image-guided percutaneous biopsy adequate for next generation sequencing (NGS), and planned to undergo core biopsy after trial registration but prior to cycle 1 day 1 of therapy; confirmation of adequacy of this biopsy material for NGS is NOT required for initiation of therapy; if elective biopsies are not being performed at the treating institution due to preparations or precautions related to coronavirus disease 2019 (COVID-19), this requirement can be waived on discussion with the trial principal investigator (PI)
* The effects of M6620 (VX-970, berzosertib), carboplatin and docetaxel on the developing human fetus are unknown. For this reason and because DNA-damage response inhibitors and chemotherapeutic agents are known to be teratogenic, men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while her partner is participating in this study, she should inform her treating physician immediately. Men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and 6 months after completion of carboplatin and M6620 (VX-970, berzosertib) administration
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Patients who have had chemotherapy or radiotherapy within 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to planned cycle 1 day 1 of study treatment; patients on an oral anti-neoplastic such as an oral hormonal agent, PARP inhibitor or oral experimental agent should discontinue >= 14 days prior to planned cycle 1 day 1 of study treatment
* Patients who have not recovered from adverse events due to prior anti-cancer therapy (i.e., have residual toxicities > grade 1), except for grade 2 anorexia, alopecia, neuropathy, and fatigue, for which resolution is not required
* Patients who are receiving any other investigational agents
* Patients with known brain metastases or leptomeningeal disease should be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to M6620 (VX-970, berzosertib) or carboplatin; (patients with allergy to docetaxel will be allowed on study, but docetaxel will be excluded from their treatment regimen)
* Subjects receiving treatment with ototoxic or nephrotoxic medications that cannot be discontinued at least 7 days before first dose of carboplatin and for the duration of the study; inadvertent or short-term use on study will not cause a subject to be ineligible; if a short course of therapy with nephrotoxic or ototoxic medication is anticipated and required, carboplatin should be discontinued until 7 days after this course is completed; patients on continuous medications that are potentially nephrotoxic who have had no evidence of nephrotoxicity from these medications at study entry are allowed to continue those medicines on trial

  * M6620 (VX-970, berzosertib) is primarily metabolized by CYP3A4; therefore, concomitant administration with strong inhibitors of CYP3A4 (e.g., ketoconazole, itraconazole, clarithromycin, ritonavir, indinavir, nelfinavir and saquinavir) or inducers of CYP3A4 (e.g. rifampin, phenytoin, carbamazepine, phenobarbital, St. John's Wort) is prohibited; because the lists of these agents are constantly changing, it is important to regularly consult a frequently-updated medical reference for a list of drugs to avoid or minimize use of; Patient Drug Information Handout and Wallet Card should be provided to patients; as part of the enrollment/informed consent procedures, the patient will be counseled on the risk of interactions with other agents, and what to do if new medications need to be prescribed or if the patient is considering a new over-the-counter medicine or herbal product
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant and nursing women are excluded from this study because they do not develop prostate cancer
* Human immunodeficiency (HIV)-positive participants with detectable viral load and/or CD4 count =< 300 are ineligible due to increased risk of lethal infections when treated with marrow-suppressive therapy; HIV-positive patients with undetectable viral loads and CD4 counts > 300, and not on interacting antiretroviral therapy may be eligible after discussing with the principal investigator
* Prior treatment with platinum-containing regimen or ATR inhibitor for prostate cancer

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2019-05-29 (Actual); Primary Completion 2021-08-10 (Actual); Study Completion 2026-04-03 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Atish D Choudhury, Principal Investigator — Dana-Farber - Harvard Cancer Center LAO
Locations (23):
- United States (23):
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - UC San Diego Moores Cancer Center, La Jolla, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - UCHealth University of Colorado Hospital, Aurora, Colorado
  - Smilow Cancer Hospital-Derby Care Center, Derby, Connecticut
  - Smilow Cancer Hospital Care Center-Fairfield, Fairfield, Connecticut
  - Smilow Cancer Hospital Care Center - Guilford, Guilford, Connecticut
  - Smilow Cancer Hospital Care Center at Saint Francis, Hartford, Connecticut
  - Smilow Cancer Center/Yale-New Haven Hospital, New Haven, Connecticut
  - Yale University, New Haven, Connecticut
  - Yale-New Haven Hospital North Haven Medical Center, North Haven, Connecticut
  - Smilow Cancer Hospital-Orange Care Center, Orange, Connecticut
  - Smilow Cancer Hospital-Torrington Care Center, Torrington, Connecticut
  - Smilow Cancer Hospital Care Center-Trumbull, Trumbull, Connecticut
  - Smilow Cancer Hospital-Waterbury Care Center, Waterbury, Connecticut
  - Smilow Cancer Hospital Care Center - Waterford, Waterford, Connecticut
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - University of Pittsburgh Cancer Institute (UPCI), Pittsburgh, Pennsylvania
  - VCU Massey Comprehensive Cancer Center, Richmond, Virginia

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 77 subjects were registered, of whom, 73 subjects underwent randomization; 4 subjects did not undergo randomization:
  1. Screen failure (n=3)
  2. Patient withdrew to pursue other treatment option (n=1)
  Patient recruitment was terminated after interim analysis showing insufficient benefit in the investigational treatment group.
Period: Overall Study
Arm/Group | Arm A (Docetaxel, Carboplatin) | Arm B (Carboplatin, Berzosertib)
Started | 37 | 36
Completed | 0 | 0
Not Completed | 37 | 36
Not completed — Never started protocol treatment | 3 | 5
Not completed — Disease progression | 11 | 16
Not completed — PSA progression | 8 | 1
Not completed — Clinical progression | 4 | 2
Not completed — Adverse Event | 5 | 4
Not completed — Intercurrent illness | 1 | 2
Not completed — Death | 1 | 1
Not completed — Withdrawal by Subject | 1 | 2
Not completed — Physician Decision | 1 | 1
Not completed — No clinical benefit | 1 | 0
Not completed — Delayed treatment for dental treatment | 1 | 0
Not completed — Difficult to maintain appointment | 0 | 1
Not completed — Protocol Violation | 0 | 1

BASELINE CHARACTERISTICS:
Population: Of 73 randomized subjects, 65 received the allocated treatment. The analysis population included the 65 subjects who received the protocol treatment: 34 in Arm A and 31 in Arm B.
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A (Docetaxel, Carboplatin) | Arm B (Carboplatin, Berzosertib) | Total
Number analyzed (Participants) | 34 | 31 | 65
Age, Continuous [Median (Inter-Quartile Range); unit: Years] — Population: The analysis population included the 65 subjects who received the protocol treatment: 34 in Arm A and 31 in Arm B.
  Years | 69 [64 to 75] | 69 [60 to 72] | 69 [62 to 72]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 34 | 31 | 65
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 3 | 6
  White | 25 | 26 | 51
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 6 | 2 | 8
Baseline Prostate-Specific Antigen (PSA) [Median (Inter-Quartile Range); unit: ng/mL] | 90 [34 to 221] | 75 [33 to 542] | 85 [34 to 375]

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate
Description: Defined by radiographic response by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 or prostate specific antigen [PSA] response (> 50% decline from baseline).
Time Frame: Radiologic measurements are performed every 3 cycles Up to 2 years. PSA measurements are performed every cycle up to 2 years
Population: The analysis population included the 65 subjects who received the protocol treatment: 34 in Arm A and 31 in Arm B.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A (Docetaxel, Carboplatin) | Arm B (Carboplatin, Berzosertib)
Number analyzed (Participants) | 34 | 31
Participants | 5 | 0

2. Secondary Outcome: Progression-free Survival (PFS)
Description: Assessed by Prostate Cancer Working Group (PCWG) 3 criteria. PFS to be estimated with the Kaplan Meier methodology. Median will be provided with 95% confidence interval.
Time Frame: From the time of randomization up to 2 years
Population: The analysis population included the 65 subjects who received the protocol treatment: 34 in Arm A and 31 in Arm B.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm A (Docetaxel, Carboplatin) | Arm B (Carboplatin, Berzosertib)
Number analyzed (Participants) | 34 | 31
Months | 2.5 [2.1 to 4.2] | 2.4 [2.1 to 3.5]

3. Secondary Outcome: Time to PSA Progression
Description: Assessed by PCWG2. PSA progression will be estimated with the Kaplan Meier methodology. Median will be provided with 95% confidence interval.
Time Frame: From the time of randomization up to 2 years
Population: The analysis population included the 65 subjects who received the protocol treatment: 34 in Arm A and 31 in Arm B.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm A (Docetaxel, Carboplatin) | Arm B (Carboplatin, Berzosertib)
Number analyzed (Participants) | 34 | 31
Months | 2.1 [1.4 to 3.6] | 1.4 [1.0 to 2.8]

4. Secondary Outcome: Radiographic Progression-free Survival (rPFS)
Description: Assessed by RECIST 1.1 for non-osseous disease and by PCWG3 for osseous disease. rPFS will be estimated with the Kaplan Meier methodology. Median will be provided with 95% confidence interval.
Time Frame: From the time of randomization up to 2 years
Population: The analysis population included the 65 subjects who received the protocol treatment: 34 in Arm A and 31 in Arm B.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm A (Docetaxel, Carboplatin) | Arm B (Carboplatin, Berzosertib)
Number analyzed (Participants) | 34 | 31
Months | 3.2 [2.1 to 5.1] | 2.6 [2.1 to 4.8]

5. Secondary Outcome: Incidence of Adverse Events
Description: Adverse events will be graded and analyzed using Common Terminology Criteria for Adverse Events (CTCAE) version 5.0.
Time Frame: Up to 2 years (from treatment initiation to 30 days after the last dose of study treatment)
Population: The analysis population included the 65 subjects who received the protocol treatment: 34 in Arm A and 31 in Arm B.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A (Docetaxel, Carboplatin) | Arm B (Carboplatin, Berzosertib)
Number analyzed (Participants) | 34 | 31
Participants | 34 | 31

6. Other Pre Specified Outcome: Overall Survival (OS)
Description: OS will be estimated with the Kaplan Meier methodology.
Time Frame: From the time of randomization up to 2 years
Population: The analysis population included the 65 subjects who received the protocol treatment: 34 in Arm A and 31 in Arm B.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm A (Docetaxel, Carboplatin) | Arm B (Carboplatin, Berzosertib)
Number analyzed (Participants) | 34 | 31
Months | 8.4 [4.5 to 12.8] | 5.7 [4.6 to 8.1]

7. Other Pre Specified Outcome: Gene Mutation Frequencies
Description: The frequency of homologous recombination (HR) deficiency detected from baseline tumor biopsy is summarized by arm at baseline.
Time Frame: At baseline
Population: Only 36 subjects had HR mutation data from baseline tumor biopsies: 22 in Arm A and 14 in Arm B.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A (Docetaxel, Carboplatin) | Arm B (Carboplatin, Berzosertib)
Number analyzed (Participants) | 22 | 14
Participants | 3 | 3

ADVERSE EVENTS:
Time Frame: From treatment initiation to 30 days after the last dose of study treatment, up to 2 years
Description: The analysis population includes 65 subjects who receive the study treatment (Arm A: 34; Arm B: 31). Adverse events are graded using Common Terminology Criteria for Adverse Events version 5.0. All-cause mortalities capture deaths within 30-days post-treatment. Serious AEs (SAE) include clinically significant AEs that are fatal, life-threatening, hospitalization-requiring, or require intervention to prevent permanent impairment; all other AEs are no-SAEs (maximum grade reported).
Arm/Group | Arm A (Docetaxel, Carboplatin) | Arm B (Carboplatin, Berzosertib)
All-Cause Mortality (participants affected / at risk) | 1/34 | 2/31
Serious Adverse Events (participants affected / at risk) | 11/34 | 14/31
Other Adverse Events (participants affected / at risk) | 34/34 | 31/31
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A (Docetaxel, Carboplatin) (N=34) | Arm B (Carboplatin, Berzosertib) (N=31)
Anemia (Blood and lymphatic system disorders) | 1 | 6
Demand Ischemia (Cardiac disorders) | 1 | 0
Myocardial Infarction (Cardiac disorders) | 1 | 0
Sinus Tachycardia (Cardiac disorders) | 0 | 1
Abdominal Pain (Gastrointestinal disorders) | 1 | 2
Ascites (Gastrointestinal disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 1 | 0
Rectal Obstruction (Gastrointestinal disorders) | 0 | 1
Rectal Pain (Gastrointestinal disorders) | 0 | 1
Death Nos (General disorders) | 1 | 0
Edema Limbs (General disorders) | 0 | 1
Fatigue (General disorders) | 2 | 0
Fever (General disorders) | 1 | 4
Gait Disturbance (General disorders) | 0 | 1
Malaise (General disorders) | 1 | 0
Pain (General disorders) | 1 | 2
Abdominal Infection (Infections and infestations) | 0 | 1
Enterocolitis Infectious (Infections and infestations) | 1 | 0
Lung Infection (Infections and infestations) | 1 | 1
Sepsis (Infections and infestations) | 0 | 2
Tooth Infection (Infections and infestations) | 0 | 1
Urinary Tract Infection (Infections and infestations) | 1 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 1
Fracture (Injury, poisoning and procedural complications) | 1 | 0
Hip Fracture (Injury, poisoning and procedural complications) | 1 | 0
Infusion Related Reaction (Injury, poisoning and procedural complications) | 1 | 0
Alanine Aminotransferase Increased (Investigations) | 1 | 0
Aspartate Aminotransferase Increased (Investigations) | 1 | 0
Blood Bilirubin Increased (Investigations) | 1 | 0
Creatinine Increased (Investigations) | 1 | 0
Neutrophil Count Decreased (Investigations) | 1 | 0
Platelet Count Decreased (Investigations) | 1 | 2
Anorexia (Metabolism and nutrition disorders) | 1 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Hypercalcemia (Metabolism and nutrition disorders) | 1 | 0
Hyperphosphatemia (Metabolism and nutrition disorders) | 0 | 1
Hypocalcemia (Metabolism and nutrition disorders) | 0 | 1
Hypokalemia (Metabolism and nutrition disorders) | 0 | 1
Hypomagnesemia (Metabolism and nutrition disorders) | 1 | 1
Back Pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Bone Pain (Musculoskeletal and connective tissue disorders) | 1 | 2
Generalized Muscle Weakness (Musculoskeletal and connective tissue disorders) | 2 | 0
Muscle Weakness Lower Limb (Musculoskeletal and connective tissue disorders) | 0 | 1
Pathologic Fracture (Musculoskeletal and connective tissue disorders) | 0 | 1
Progressive Disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Tumor Pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Encephalophathy (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 1 | 0
Spinal Cord Compression (Nervous system disorders) | 0 | 1
Confusion (Psychiatric disorders) | 1 | 0
Acute Kidney Injury (Renal and urinary disorders) | 0 | 1
Hematuria (Renal and urinary disorders) | 1 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hypotension (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A (Docetaxel, Carboplatin) (N=34) | Arm B (Carboplatin, Berzosertib) (N=31)
Anemia (Blood and lymphatic system disorders) | 18 | 20
Platelet Count Decreased (Investigations) | 16 | 20
Fatigue (General disorders) | 14 | 15
Nausea (Gastrointestinal disorders) | 11 | 13
Constipation (Gastrointestinal disorders) | 10 | 14
Aspartate Aminotransferase Increased (Investigations) | 9 | 6
Anorexia (Metabolism and nutrition disorders) | 9 | 11
Diarrhea (Gastrointestinal disorders) | 7 | 6
Neutrophil Count Decreased (Investigations) | 7 | 7
Abdominal Pain (Gastrointestinal disorders) | 6 | 3
Hypocalcemia (Metabolism and nutrition disorders) | 6 | 7
Dysgeusia (Nervous system disorders) | 6 | 4
Alkaline Phosphatase Increased (Investigations) | 5 | 5
White Blood Cell Decreased (Investigations) | 5 | 11
Hypoalbuminemia (Metabolism and nutrition disorders) | 5 | 2
Hematuria (Renal and urinary disorders) | 5 | 5
Vomiting (Gastrointestinal disorders) | 4 | 5
Edema Limbs (General disorders) | 4 | 1
Alanine Aminotransferase Increased (Investigations) | 4 | 3
Blood Lactate Dehydrogenase Increased (Investigations) | 4 | 0
Lymphocyte Count Decreased (Investigations) | 4 | 7
Weight Loss (Investigations) | 4 | 7
Hyponatremia (Metabolism and nutrition disorders) | 4 | 6
Hypophosphatemia (Metabolism and nutrition disorders) | 4 | 4
Bone Pain (Musculoskeletal and connective tissue disorders) | 4 | 4
Peripheral Sensory Neuropathy (Nervous system disorders) | 4 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 4 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 4 | 10
Watering Eyes (Eye disorders) | 3 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 3 | 5
Hypokalemia (Metabolism and nutrition disorders) | 3 | 6
Back Pain (Musculoskeletal and connective tissue disorders) | 3 | 6
Tremor (Nervous system disorders) | 3 | 0
Hypotension (Vascular disorders) | 3 | 4
Sinus Tachycardia (Cardiac disorders) | 2 | 4
Chills (General disorders) | 2 | 3
Fever (General disorders) | 2 | 8
Generalized Edema (General disorders) | 2 | 1
Pain (General disorders) | 2 | 4
Thrush (Infections and infestations) | 2 | 0
Upper Respiratory Infection (Infections and infestations) | 2 | 1
Urinary Tract Infection (Infections and infestations) | 2 | 4
Creatinine Increased (Investigations) | 2 | 7
Dehydration (Metabolism and nutrition disorders) | 2 | 1
Hypomagnesemia (Metabolism and nutrition disorders) | 2 | 6
Generalized Muscle Weakness (Musculoskeletal and connective tissue disorders) | 2 | 6
Dizziness (Nervous system disorders) | 2 | 8
Headache (Nervous system disorders) | 2 | 3
Paresthesia (Nervous system disorders) | 2 | 3
Thromboembolic Event (Vascular disorders) | 2 | 3
Tinnitus (Ear and labyrinth disorders) | 1 | 2
Bruising (Injury, poisoning and procedural complications) | 1 | 2
Infusion Related Reaction (Injury, poisoning and procedural complications) | 1 | 2
LDH increase (Investigations) | 1 | 3
Muscle Cramp (Musculoskeletal and connective tissue disorders) | 1 | 3
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 2
Neck Pain (Musculoskeletal and connective tissue disorders) | 1 | 2
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 1 | 4
Depression (Psychiatric disorders) | 1 | 2
Pelvic Pain (Reproductive system and breast disorders) | 1 | 3
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 2
Hot Flashes (Vascular disorders) | 1 | 2
Hypertension (Vascular disorders) | 1 | 3
Dyspepsia (Gastrointestinal disorders) | 0 | 2
Gastroparesis (Gastrointestinal disorders) | 0 | 2
Hyperkalemia (Metabolism and nutrition disorders) | 0 | 2
Hyperphosphatemia (Metabolism and nutrition disorders) | 0 | 2
Flank Pain (Musculoskeletal and connective tissue disorders) | 0 | 2
Muscle Weakness Lower Limb (Musculoskeletal and connective tissue disorders) | 0 | 3
Proteinuria (Renal and urinary disorders) | 0 | 2
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Rash Maculo-Papular (Skin and subcutaneous tissue disorders) | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-08-24): https://cdn.clinicaltrials.gov/large-docs/69/NCT03517969/Prot_SAP_000.pdf
  • Informed Consent Form (2024-08-24): https://cdn.clinicaltrials.gov/large-docs/69/NCT03517969/ICF_002.pdf